CLINICAL TRIAL: NCT01982357
Title: Measurement of Neonatal Microvascular Hemodynamics Using Non-invasive Optical Technologies
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Omid Fathi, M.D., Pediatrics, University of California, Irvine
Other Study IDs: 20139505
Record Dates: First submitted 2013-11-05; First posted 2013-11-13 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases | interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- premature infant: Laser Speckle Imaging and Diffuse Optical Spectroscopy
  Interventions: Device: Laser Speckle Imaging and Diffuse Optical Spectroscopy

INTERVENTIONS:
Device: Laser Speckle Imaging and Diffuse Optical Spectroscopy — Laser Speckle Imaging and Diffuse Optical Spectroscopy

SUMMARY:
Alterations to microvascular blood flow in premature infants, are known to contribute to several major disease entities.

The optically-measured tissue blood flow, to determine tissue perfusion that can be use to detect blood loss.

DETAILED DESCRIPTION:
The researchers want to use optical technologies to non-invasively detect blood flow that can tell the onset of blood loss. The research can measure blood flow in stable premature infants in the Neonatal Intensive Care Unit over the duration of several weeks.

The technologies are Laser Speckle Imaging and Diffuse Optical Spectroscopy.

Laser Speckle Imaging non-contact imaging technology, is sensitive to blood flow in superficial tissues. Diffuse Optical Spectroscopy, a probe-based contact technology like pulse oximetry, measures hemoglobin concentrations and states deeper below the skin surface.

ELIGIBILITY:
Inclusion Criteria:

* premature infants born or transferred to neonatal intensive care unit with a gestational age of 28-35 weeks

Exclusion Criteria:

* NONE premature infants born or transferred to neonatal intensive care unit

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study population will be selected from University of California Irvine Medical Center at Neonate Intensive Care Unit
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Normal Blood flow in premature infant | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Omid Fathi, MD, Principal Investigator — Beckman Laser Institute, UCI; Bernard Choi, PhD, Study Director — Beckman Laser Institute, UCI
Locations (1):
- UCIMC, Orange, California, United States